CLINICAL TRIAL: NCT00770068
Title: Seasonality of Depression and Airborne Allergens
Brief Title: Examining the Link Between Depression and Seasonal Allergies
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Teodor Postolache, Professor, University of Maryland, Baltimore
Other Study IDs: R21MH075891 (NIH); R21MH075891 (NIH); H26191; DATR A2-AID
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Depression
Keywords: Mood Disorders; Major Depressive Disorder; Bipolar Disorder; Tree Pollen; Ragweed Pollen; Rhinitis; Allergic; Seasonal; Allergens
MeSH Terms: conditions — Depression; Mood Disorders; Depressive Disorder, Major; Bipolar Disorder; Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental group: All participants testing positive for tree and ragweed pollen allergies, as determined by levels of immunoglobulin E (IgE) antibodies
- Control group: All participants testing negative for tree and ragweed pollen allergies, as determined by levels of IgE antibodies

SUMMARY:
This study will examine whether spring and fall seasonal depression in individuals with high sensitivity to pollen is linked to seasonal increases in tree and ragweed pollen.

DETAILED DESCRIPTION:
Those who suffer from depression have their normal lives interrupted by symptoms such as persistent sad thoughts, inability to feel pleasure, and potential suicide. Suicide and depression peak in the spring and fall. Worsening of depression, admission to a hospital for depression and bipolar depression, and use of electroconvulsive therapy for treatment of depression all peak in the spring. Although seasonal affective disorder (SAD), in which depression corresponds with seasonal changes, is commonly associated with the winter subtype, SAD is actually more prevalent as the spring subtype.

Allergies, which also peak in the spring and fall, have been linked to depression. Allergic reactions release cytokines, which are proteins that mediate the immune system response when a foreign substance enters the body. Previous studies have found both that an increase in cytokines in otherwise healthy individuals causes depressive symptoms and that cytokines cause the chemical tryptophan (TRP) to switch from producing serotonin, a neurotransmitter associated with feelings of well-being, to producing kynurenine (KYN), a potentially toxic chemical. To determine whether and to what extent allergies are linked to depression, this study will compare depression levels of participants with and without allergies before and during peak times for seasonal allergies. Results from this study may be used in further research to examine the effects of allergy prevention on depression.

Participants in this study will meet with researchers three times. At the first visit, they will be screened for allergies and give their demographic information. The timing of the second and third visits will depend on each participant's allergies. Those with spring allergies will be tested before and then during the spring allergy season. Those with fall allergies or with no allergies will be tested before and then during the fall allergy season. On the second and third visits questionnaires and clinical interviews will assess depression symptoms, and blood tests will be performed to measure chemical levels of cytokines, TRP, and KYN. During these visits participants will also be asked to complete a sleep log for 1 week. This will entail describing their sleep, activity, caffeine consumption, alcohol consumption, and use of sleep medications. A subgroup will wear an Actiwatch device, which electronically monitors sleep and wakefulness cycles, for 1 week, 24 hours a day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder or bipolar disorder

Exclusion Criteria:

* Pregnancy or intention to become pregnant within the duration of the study
* Dependence on alcohol, cocaine, stimulants, benzodiazepines, marijuana, or opiates
* Major medical illness, including cancer, hepatitis, and autoimmune disease
* A winter subtype of seasonal affective disorder
* Diagnosis of psychotic disorder
* Positive result in Phadiatop allergy test, but negative result in tree or ragweed pollen IgE test

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A community sample will be recruited via local press and radio advertising. Referrals from mental health providers will be used to supplement this population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-07-15; Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression-Seasonal Affective Disorder Version (SIGH-SAD) | Measured before and then during the peak fall or spring pollen period

SECONDARY OUTCOMES:
Hypomania Interview Guide (HIGH-SAD) | Measured before and then during the peak fall or spring pollen period
Burns Anxiety Inventory | Measured before and then during the peak fall or spring pollen period
Buss Aggression Questionnaire | Measured before and then during the peak fall or spring pollen period
Allergy Symptom Severity Assessment (ASSA) Questionnaire | Measured before and then during the peak fall or spring pollen period
Serum cytokine, tryptophan (TRP), and kynurenine (KYN) concentrations | Measured before and then during the peak fall or spring pollen period
Nasal secretion test | Measured before and then during the peak fall or spring pollen period
Sleep logs | Measured over 1 week during pre- or post-pollen and peak pollen period
Actiwatch | Measured after the pre-pollen and peak pollen visits for 24 hours a day for 1 week
Beck Depression Inventory II (BDI-II) | Measured during the peak pollen period
Pittsburgh Sleep Quality Index (PSQI) | Measured during the peak pollen period

CONTACTS AND LOCATIONS:
Overall Officials: Teodor T. Postolache, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - National Center for the Treatment of Phobias, Anxiety, and Depression, Washington D.C., District of Columbia
  - University of Maryland, Baltimore, Maryland

REFERENCES:
- [Background] Manalai P, Hamilton RG, Langenberg P, Kosisky SE, Lapidus M, Sleemi A, Scrandis D, Cabassa JA, Rogers CA, Regenold WT, Dickerson F, Vittone BJ, Guzman A, Balis T, Tonelli LH, Postolache TT. Pollen-specific immunoglobulin E positivity is associated with worsening of depression scores in bipolar disorder patients during high pollen season. Bipolar Disord. 2012 Feb;14(1):90-8. doi: 10.1111/j.1399-5618.2012.00983.x. PMID 22329476
- [Result] Postolache TT, Lapidus M, Sander ER, Langenberg P, Hamilton RG, Soriano JJ, McDonald JS, Furst N, Bai J, Scrandis DA, Cabassa JA, Stiller JW, Balis T, Guzman A, Togias A, Tonelli LH. Changes in allergy symptoms and depression scores are positively correlated in patients with recurrent mood disorders exposed to seasonal peaks in aeroallergens. ScientificWorldJournal. 2007 Dec 17;7:1968-77. doi: 10.1100/tsw.2007.286. PMID 18167612